CLINICAL TRIAL: NCT05791695
Title: A US Real-World Evidence Study of the Incidence of Intraocular Inflammation and Suspected Endophthalmitis Among Patients Treated With Aflibercept, Vial and Pre-filled Syringe, 2014-2022
Brief Title: A Study of the Incidence of Intraocular Inflammation and Suspected Endophthalmitis Among Patients Treated With Aflibercept, Vial and Pre-filled Syringe, 2014-2022
Status: Completed | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: VGFTe-OD-2222
Record Dates: First submitted 2023-02-27; First posted 2023-03-30 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-10

CONDITIONS: Intraocular Inflammation; Suspected Endophthalmitis
Keywords: Age-related macular degeneration; Anti-vascular endothelial growth factor; Diabetic macular edema; Diabetic retinopathy; Endophthalmitis; Intraocular inflammation; Retinal vein occlusion; Vascular endothelial growth factor
MeSH Terms: conditions — Uveitis; Macular Degeneration; Diabetic Retinopathy; Endophthalmitis; Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Patients: Patients ≥ 18 years who have received one or more injections of aflibercept during the study period
  Interventions: Other: Non Applicable

INTERVENTIONS:
Other: Non Applicable — No study-specific interventions for this observational study.

SUMMARY:
Specific study objectives include:

* To describe patient and provider characteristics for aflibercept patients and aflibercept user injections by aflibercept dispensing device, overall, and stratified by time (quarterly, annually).
* To estimate the annual and quarterly incidence of intraocular inflammation (IOI) and suspected endophthalmitis for aflibercept user injections by aflibercept dispensing device.

Secondary objectives

• To estimate the annual incidence of IOI and suspected endophthalmitis for aflibercept user injections by dispensing device, stratified by indication for use, history of IOI, and provider characteristics.

DETAILED DESCRIPTION:
This study is entirely descriptive using secondary data from the Vestrum Health Retina Treatment and Outcomes database.

ELIGIBILITY:
Inclusion Criteria for a Treatment Episode:

1. Must have received one or more injections of aflibercept, regardless of indication, between 01Jan2014 to 30Apr2022
2. Patients must have at least one eligible treatment episode a. Specification of laterality of aflibercept injection (left or right eye or both) for treatment episode

Exclusion Criteria for a Treatment Episode:

1. A post-operative follow-up visit for any ocular surgery (excluding vitrectomy), within +/-28 days of aflibercept injection, as defined in the protocol
2. Active steroid treatment, defined as steroid treatment (topical or intravitreal) on the date of aflibercept injection. This criterion is limited to date of aflibercept injection since steroids may be used to treat IOIs.
3. Any treatment episode where a patient eye receives >1 (or an unknown) anti-VEGF injection on the index date (date of aflibercept injection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study period will span from 01 Jan 2014 (earliest complete data available) to 28 May 2022 (or most current data available). The study will include patients ≥18 years of age in Vestrum who have received one or more injections of aflibercept, regardless of indication, between 01 Jan 2014 to 30 Apr 2022 (one month look forward required). Patients must have at least one eligible treatment episode (defined as aflibercept injection followed by 28-day exposed period after injection) to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 155413 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Frequency of patients receiving aflibercept injections | End of Study, Approximately 8 Years
Frequency of aflibercept injections by ophthalmic delivery mechanism | End of Study, Approximately 8 Years
  Ophthalmic delivery mechanism defined as prefilled syringe (PFS) and vial
Incidence of Intraocular inflammation (IOI) | End of Study, Approximately 8 Years
  Incidence will be defined as the number of events during the at-risk period divided by the total number of injections, identified using international classification of diseases (ICD-9 and ICD-10) diagnosis codes.
Incidence of Intraocular inflammation (IOI) by ophthalmic delivery mechanism | End of Study, Approximately 8 Years
  Incidence will be defined as the number of events during the at-risk period divided by the total number of injections, identified using international classification of diseases (ICD-9 and ICD-10) diagnosis codes.
  Ophthalmic delivery mechanism defined as prefilled syringe (PFS) and vial
Incidence of suspected endophthalmitis | End of Study, Approximately 8 Years
  Incidence will be defined as the number of events during the at-risk period divided by the total number of injections, identified using international classification of diseases (ICD-9 and ICD-10) diagnosis codes.
Incidence of suspected endophthalmitis by ophthalmic delivery mechanism | End of Study, Approximately 8 Years
  Incidence will be defined as the number of events during the at-risk period divided by the total number of injections, identified using international classification of diseases (ICD-9 and ICD-10) diagnosis codes.
  Ophthalmic delivery mechanism defined as prefilled syringe (PFS) and vial

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Research Site, Tarrytown, New York, United States

IPD SHARING:
Plan to Share IPD: No